CLINICAL TRIAL: NCT03461185
Title: Anti-angiogenesis Combine With EGFR-TKI in Advanced Non-squamous Non Small Cell Cancer
Brief Title: Anti-angiogenesis Combine With EGFR-TKI in Advanced Non-squamous Non Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xinqiao Hospital of Chongqing (Other)
Responsible Party: Principal Investigator, Zhengtang Chen, Xinqiao Hospital of Chongqing, Xinqiao Hospital of Chongqing
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: xinqiao2018001
Record Dates: First submitted 2018-03-04; First posted 2018-03-09 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Angiogenesis Inhibitors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EGFR-TKI plus anti-angiogenesis (Experimental): EGFR-TKI(erlotinib or gefitinib) plus anti-angiogenesis(endostatin or apatinib or anlotinib)
  Interventions: Drug: EGFR-TK Inhibitor; Drug: Anti-Angiogenic Drugs
- EGFR-TKI (Active Comparator): EGFR-TKI(erlotinib or gefitinib)
  Interventions: Drug: EGFR-TK Inhibitor

INTERVENTIONS:
Drug: EGFR-TK Inhibitor — EGFR-TKIs include but are not limited erlotinib, gefitinib
Drug: Anti-Angiogenic Drugs — Anti-Angiogenic Drugs contain endostatin, apatinib and anlotinib
  Arms: EGFR-TKI plus anti-angiogenesis

SUMMARY:
Epidermal growth factor receptor Tyrosine kinase inhibitor (EGFR TKI) have been approved to treat NSCLC harboring EGFR mutation as first-line therapy. However, the acquired resistance of EGFR-TKI is a common and severe problem.The study explore the superiority of anti-angiogenesis drugs (Apatinib, endostatin, anlotinib) plus EGFR TKI versus single EGFR-TKI.

DETAILED DESCRIPTION:
Non-small-cell lung cancer (NSCLC) is the leading cause from cancer in China. Epidermal growth factor receptor Tyrosine kinase inhibitor (EGFR TKI) have been approved to treat NSCLC harboring EGFR mutation as first-line therapy. However, a large proportion of patients would become acquired resistant of EGFR-TKI after about one year although initially sensitivity. Anti-angiogenesis therapy plus EGFR-TKI has been demonstrated valid and safe in NSCLC patients. Apatinib, endostatin, anlotinib belong to anti-angiogenesis drugs and can inhibit tumor growth. In this study, we plan to recruit NSCLC patients who are assessed as stable disease ( according to RECIST) under treatment of EGFR-TKI. Then, these patients would be divided into two groups: single EGFR-TKI or EGFR-TKI plus anti-angiogenesis drugs. Progression free survival, overall survival and safety are our evaluation events.

ELIGIBILITY:
Inclusion Criteria:

1. Aged from 18 to 75 years (18 and 75 years are included)Obtain of informed consent.
2. Histologically or cytologically confirmed, inoperable, recurrence or metastasis advanced non-small cell lung cancer (TNM Stage ⅢB or stage Ⅳ), took EGFR-TKI longer than 2 months and appeared Stable disease.
3. At least one measurable lesion (helical CT scan long diameter ≥10mm, meet the requirements of the standard Response Evaluation Criteria In Solid Tumors（RESCIST） version 1.1).
4. Eastern Cooperative Oncology Group（ECOG）Performance Status（PS） :0-2.
5. Life expectancy ≥12 weeks.
6. Adequate bone marrow reserve and organ function as follows:

   * Absolute neutrophils count (ANC) ≥1.5 x 10 to the 9th power/L (band neutrophil and segmented neutrophil), platelets > 100 x 10 to the 9th power/L and Hb≥90g/L.

     * Hepatic: total bilirubin less than or equal to 1.5 times upper limit of normal (ULN).

       * Alkaline phosphatase (AP), alanine transaminase (ALT) and aspartate transaminase (AST) less than or equal to 3.0 times ULN (or less than or equal to 5 times ULN in case of known liver involvement.

         * Renal: Serum Creatinine less than or equal to 1.25 times upper limit of normal (ULN).
7. Females of child-bearing potential must have negative serum pregnancy test. Sexually active males and females (of childbearing potential) willing to practice contraception during the study.

Exclusion Criteria:

1. Do not meet the above criteria.
2. Unhealed toxicity of prior anti-cancer treatment (CTCAE Level 1) or surgery. Uncontrolled hypertension (systolic ≥140mmHg and/or diastolic ≥90mmHg after medication treatment).
3. Clinical uncontrolled active infection, such as acute pneumonia, active hepatitis B or C (prior hepatitis B history, despite medication treatment control or not, HBV DNA≥500copies or ≥100IU/ml), etc.
4. Arterial thrombosis or venous thrombosis in 6 months, or disposition evidence of thrombosis/bleeding in 2 month (despite severity), hemoptysis in 2 weeks (bright red blood, 1/2 teaspoon).
5. Stroke or transient ischemic attack (TIA) in 12 month. Unhealed skin lesions, surgical site, injuries, severe mucous membrane ulcer or bone fracture.
6. Cardiac function evaluation: LVEF <50%, a recent history of MI in 6 months, severe/unstable angina or coronary bypass surgery, or cardiac insufficiency ≥ NYHA 2.
7. Prior other malignant disease in 5 years.
8. Recent active digestive disease such as duodenal ulcers, ulcerative colitis, ileus, ect., intestinal perforation, intestine fistula, or other conditions may lead to gastrointestinal bleeding or perforation which regimented at investigators' discretion.
9. Difficulty swallowing or known malabsorption.
10. A history of organ transplantation and long-term immunosuppressive medication.
11. Take part in new drug clinical trials within one month or taking part in a trial now.
12. Pregnant or lactating woman.
13. Other conditions regimented at investigators' discretion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2019-08-30 (Estimated); Study Completion 2020-02-20 (Estimated)

PRIMARY OUTCOMES:
Progression free survival(PFS) | 24 months
  PFS is evaluated in 24 months since the treatment begin

SECONDARY OUTCOMES:
Overall survival (0S) | 24 months
  OS is evaluated in 24 months since the treatment begin

CONTACTS AND LOCATIONS:
Locations (1):
- XinQiao Hospital, Chongqing, Chongqing Municipality, China